CLINICAL TRIAL: NCT04638036
Title: Fluorescence Molecular Endoscopy and Molecular Fluorescence-guided Surgery of Locally Advanced Rectal Cancer Using Cetuximab-IRDye800CW: a Single-center Feasibility and Safety Study
Brief Title: Fluorescence Molecular Endoscopy and Molecular Fluorescence-guided Surgery in Locally Advanced Rectal Cancer
Acronym: TRACT-II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL61406.042.17
Record Dates: First submitted 2020-11-03; First posted 2020-11-20 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIR endoscopy and surgery with cetuximab-IRDye800CW (Experimental): In this non-randomized, non-blinded, prospective, feasibility study, cetuximab-IRDye800CW will be administered to a total of 15 patients with proven locally advanced rectal cancer
  Interventions: Drug: Cetuximab-IRDye800; Device: Fluorescent molecular endoscopy and surgery

INTERVENTIONS:
Drug: Cetuximab-IRDye800 — Intravenous administration of a pre-dose of 75 mg unlabeled Cetuximab followed by 15 mg Cetuximab-IRDye800 prior to the study procedures
  Other Names: Tracer administration
Device: Fluorescent molecular endoscopy and surgery — A flexible fluorescence fiber-bundle is attached to a fluorescence camera platform to enable the detection of fluorescence signals. The fluorescence fiber-probe can be inserted through the standard working channel of the standard clinical endoscope for fluorescent endoscopy. Fluorescence imaging will be performed post the chemoradiotherapy.

SUMMARY:
Treatment of patients with locally advanced rectal cancer (LARC) is multidisciplinary and consists of neoadjuvant chemoradiotherapy (nCRT) followed by surgical removal of the rectal tumor and potentially tumor positive lymph nodes.

1. After surgery, in 15 to 27% of patients that received nCRT no tumor cells can be detected during histopathological examination. In today's clinical practice, all of these patients with a pathological complete response (pCR) are operated upon, with substantial morbidity and mortality. The 5-year survival is 83.3% for patients with a pCR, and 65.6% for those without pCR. Response after nCRT is currently evaluated using magnetic resonance imaging (MRI). However, as MRI cannot differentiate between molecular characteristics of tissue, prediction of treatment response can be inaccurate. In patients with a potential cCR on MRI, additionally a high-definition white-light (HD-WL) endoscopy is performed with biopsies of the previous tumor location. If both MRI and HD-WL endoscopy confirm a potential cCR, patients can also be treated with a watch-and-wait approach, including frequent follow-up with HD-WL endoscopy and MRI. This potentially prevents extensive surgical procedures for patients in which this is not required. However, MRI and HD-WL endoscopy often remain insufficient for identification of cCR. Therefore, novel imaging methods are needed for accurate prediction of treatment response in order to select patients. The investigators believe fluorescence molecular endoscopy (FME) could be a promising technique for evaluation of treatment response.
2. During surgery, tumor-negative resection margins are of great prognostic value. Currently, surgeons rely on visual and tactile inspection for differentiation between malignant and healthy tissue. When in doubt, a frozen section can be obtained, which is time consuming and poses a high risk of sampling error. However, 14.7% of patients still have tumor-positive resection margins, increasing the risk of local recurrence and worsening outcome. Therefore, there is a need for novel imaging techniques that can be used intraoperatively to improve margin assessment. The investigators believe molecular fluorescence-guided surgery (MFGS) could be a promising technique for evaluation of resection margins.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced rectal cancer, in multi-disciplinary colorectal oncology meeting agreed on long course neoadjuvant chemoradiotherapy, followed by surgical removal of the primary tumor;
* Clinical suspicion of residual tumor after neoadjuvant chemoradiotherapy;
* Age ≥ 18 years;
* Written informed consent.

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent;
* Concurrent uncontrolled medical conditions;
* Pregnancy or breast feeding. A negative pregnancy test must be available for women of childbearing potential (i.e. premenopausal women with intact reproductive organs and women less than two years after menopause);
* Received an investigational drug within 30 days prior to the dose of cetuximab- IRDye800CW;
* History of infusion reactions to cetuximab or other monoclonal antibodies;
* Had within 6 months prior to enrollment: myocardial infarction, cerebrovascular accident, uncontrolled cardiac heart failure, significant liver disease, unstable angina pectoris;
* Patients receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents;
* Evidence of QT prolongation on an ECG made within three months prior to inclusion (greater than 440 ms in males or greater than 450 ms in females);
* Magnesium, potassium and calcium deviations that might lead to cardiac rhythm (grade II or higher deviations by CTCAE), determined within three months prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2023-05-21 (Actual)

PRIMARY OUTCOMES:
Safety of molecular fluorescence endoscopy using Cetuximab-800CW | up to 3 months
  Number of participants with treatment-related (serious) adverse events
Safety of molecular fluorescence-guided surgery using Cetuximab-800CW | up to 3 months
  Number of participants with treatment-related (serious) adverse events
Feasibility of molecular fluorescence endoscopy using Cetuximab-800CW | up to 3 months
  Feasibility will be evaluated by assessing real-time during endoscopy whether fluorescence can be visualized and by taking images during fluorescence molecular endoscopy. Thereafter the fluorescence intensity using the raw data will be measured and a tumor-to-background ratio will be calculated.
Feasibility of molecular fluorescence-guided surgery using Cetuximab-800CW | up to 3 months
  Feasibility will be evaluated by assessing whether fluorescence can be detected in the resection margins and on the specimen. Thereafter the fluorescence intensity using the raw data will be measured and a tumor-to-background ratio will be calculated.

SECONDARY OUTCOMES:
Quantifcation of the fluorescent signals | up to 3 months
  To quantify fluorescence signals in vivo and ex vivo using multi-diameter single-fiber reflectance, single-fiber fluorescence (MDSFR/SFF) spectroscopy measurements
Correlation of the fluorescent signal to histopathology and immunohistochemistry | up to 3 months
  To correlate and validate fluorescence signals detected in vivo with ex vivo histopathology and immunohistochemistry
Evaluation of the distribution of Cetuximab-IRDye800CW | up to 3 months
  To evaluate the distribution of cetuximab-IRDye800CW on a microscopic level using fluorescence microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands